CLINICAL TRIAL: NCT00363129
Title: The Use of Vitamin E for Prevention of Chemotherapy Induced Peripheral Neuropathy: A Phase III Double-Blind Placebo Controlled Study
Brief Title: Vitamin E in Preventing Peripheral Neuropathy Caused by Chemotherapy in Patients Receiving Chemotherapy for Cancer
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Alliance for Clinical Trials in Oncology (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: NCCTG-N05C3; NCI-2011-01712 (Registry Identifier: CTRP (Clinical Trials Reporting System)); CDR0000491071 (Registry Identifier: PDQ (Physician Data Query))
Record Dates: First submitted 2006-08-10; First posted 2006-08-15 (Estimated); Results first posted 2014-08-08 (Estimated); Last update posted 2016-07-06 (Estimated); Status verified 2016-07

CONDITIONS: Neurotoxicity; Unspecified Adult Solid Tumor, Protocol Specific
Keywords: neurotoxicity; unspecified adult solid tumor, protocol specific
MeSH Terms: conditions — Neurotoxicity Syndromes | interventions — Vitamin E

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Arm I (Experimental): Patients receive oral vitamin E twice daily beginning within 4 days of the start of chemotherapy course 1 and continuing until 1 month after completion of chemotherapy.
  Interventions: Dietary Supplement: vitamin E
- Arm II (Placebo Comparator): Patients receive oral placebo twice daily beginning within 4 days of the start of chemotherapy course 1 and continuing until 1 month after completion of chemotherapy.
  Interventions: Other: placebo

INTERVENTIONS:
Dietary Supplement: vitamin E — Given orally
  Arms: Arm I
Other: placebo — Given orally
  Arms: Arm II

SUMMARY:
RATIONALE: Vitamin E may prevent peripheral neuropathy caused by chemotherapy in patients with cancer. It is not yet known whether vitamin E is more effective than a placebo in preventing peripheral neuropathy caused by chemotherapy in patients receiving chemotherapy for cancer.

PURPOSE: This randomized phase III trial is studying vitamin E to see how well it works compared with placebo in preventing peripheral neuropathy caused by chemotherapy in patients receiving chemotherapy for cancer.

DETAILED DESCRIPTION:
OUTLINE: This is a randomized, double-blind, placebo-controlled, multicenter study. Patients are stratified according to type of chemotherapy (taxane vs cisplatin vs carboplatin vs oxaliplatin vs combination), age (≤ 50 years vs > 50 years), and gender. Patients are randomized to 1 of 2 treatment arms.

OBJECTIVES:

Primary

* Compare the incidence of chemotherapy-induced sensory peripheral neuropathy ≥ grade 2 in patients undergoing curative neurotoxic chemotherapy for cancer treated with vitamin E vs placebo.

Secondary

* Compare the proportion of patients requiring dose reductions of chemotherapy secondary to sensory peripheral neuropathy.
* Compare the proportion of patients stopping chemotherapy before treatment is complete secondary to sensory peripheral neuropathy.
* Assess the toxicity of vitamin E in these patients.

After completion of study treatment, patients are followed at 6 months.

ELIGIBILITY:
Required Characteristics:

1. Scheduled to undergo curative-intent adjuvant treatment with neurotoxic chemotherapy. Patients must have had his/her tumor removed, but may have microscopic residual disease, or residual margin involvement and still be eligible.

   The patient's chemotherapy regimen must include one or more of the following neurotoxic chemotherapeutic agents: taxanes (paclitaxel, docetaxel); platinum compounds (cisplatin, carboplatin, oxaliplatin)-(oxaliplatin patients should preferentially be enrolled in protocol N04C7 while it is available).
2. ≥ 18 years of age
3. Ability to sign informed consent and understand the nature of a placebo-controlled trial
4. ECOG Performance Status (PS) of 0, 1, or 2 e.g.
5. Ability to complete questionnaire(s) by themselves or with assistance
6. Life expectancy ≥ 6 months

Contraindications:

1. Undergoing chemotherapy for palliative care
2. Pre-existing history of peripheral neuropathy due to any cause (diabetes, alcohol, toxin, hereditary, etc).
3. Prior treatment with neurotoxic chemotherapy (exception: Patient started neurotoxic chemotherapy ≤ 4 days of starting vitamin E on this study and has not been treated previously with other neurotoxic chemotherapy agents).
4. Taking regular opioid-containing medications. (Exception: opioids, given for the short term treatment of chemotherapy-induced myalgias or arthralgias caused by taxanes are permitted.)
5. Concurrent treatment with anticonvulsants, tricyclic antidepressants, or other neuropathic pain medications agents such as carbamazepine, phenytoin, valproic acid, gabapentin, lamotrigine, topical lidocaine patch, capsaicin cream, etc.
6. History of coronary artery disease (i.e. MI, PTCA, or CABG ≤ 5 years or diagnosis of congestive heart failure of any NY heart class I-IV) Valve replacements are permitted as long as patient has fully recovered from the surgery.
7. Other medical conditions, which in the opinion of the treating physician/allied health professional would make this protocol unreasonably hazardous for the patient.
8. Vitamin E supplementation for any reason ≤ 7 days prior to randomization. (Exception:

   one multivitamin per day that contains ≤ 100 IU [mg] of Vitamin E, will be permitted.)
9. Any of the following: pregnant women, nursing women and men or women of childbearing potential who are unwilling to employ adequate contraception
10. Taking anticoagulant medication (i.e. coumadin, low molecular weight heparin (LMWH), or platelet aggregation inhibitors such as clopidgrel or aspirin) with the exception that 1 mg/day of coumadin for central line maintenance is allowed.
11. Diagnosed diabetes requiring insulin or oral hypoglycemic medications
12. Head or neck cancers
13. Scheduled to undergo radiation therapy while on study
14. History of hemorrhagic stroke
15. Patients receiving neo-adjuvant therapy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 207 (Actual)
Dates: Start 2006-12; Primary Completion 2010-12 (Actual); Study Completion 2014-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Lisa Kottschade, RN, MSN, CNP, Study Chair — Mayo Clinic
Locations (69):
- United States (69):
  - St. Joseph Medical Center, Bloomington, Illinois
  - Graham Hospital, Canton, Illinois
  - Memorial Hospital, Carthage, Illinois
  - Eureka Community Hospital, Eureka, Illinois
  - Galesburg Clinic, PC, Galesburg, Illinois
  - Galesburg Cottage Hospital, Galesburg, Illinois
  - Mason District Hospital, Havana, Illinois
  - Hopedale Medical Complex, Hopedale, Illinois
  - Joliet Oncology-Hematology Associates, Limited - West, Joliet, Illinois
  - Kewanee Hospital, Kewanee, Illinois
  - BroMenn Regional Medical Center, Normal, Illinois
  - Community Cancer Center, Normal, Illinois
  - Community Hospital of Ottawa, Ottawa, Illinois
  - Oncology Hematology Associates of Central Illinois, PC - Ottawa, Ottawa, Illinois
  - CCOP - Illinois Oncology Research Association, Peoria, Illinois
  - Oncology Hematology Associates of Central Illinois, PC - Peoria, Peoria, Illinois
  - Perry Memorial Hospital, Princeton, Illinois
  - Carle Cancer Center at Carle Foundation Hospital, Urbana, Illinois
  - CCOP - Carle Cancer Center, Urbana, Illinois
  - Saint Anthony Memorial Health Centers, Michigan City, Indiana
  - McCreery Cancer Center at Ottumwa Regional, Ottumwa, Iowa
  - Siouxland Hematology-Oncology Associates, LLP, Sioux City, Iowa
  - St. Luke's Regional Medical Center, Sioux City, Iowa
  - Saint Joseph Mercy Cancer Center, Ann Arbor, Michigan
  - CCOP - Michigan Cancer Research Consortium, Ann Arbor, Michigan
  - Oakwood Cancer Center at Oakwood Hospital and Medical Center, Dearborn, Michigan
  - Genesys Hurley Cancer Institute, Flint, Michigan
  - Van Elslander Cancer Center at St. John Hospital and Medical Center, Grosse Pointe Woods, Michigan
  - Foote Memorial Hospital, Jackson, Michigan
  - Sparrow Regional Cancer Center, Lansing, Michigan
  - Seton Cancer Institute at Saint Mary's - Saginaw, Saginaw, Michigan
  - St. John Macomb Hospital, Warren, Michigan
  - Fairview Ridges Hospital, Burnsville, Minnesota
  - Mercy and Unity Cancer Center at Mercy Hospital, Coon Rapids, Minnesota
  - Fairview Southdale Hospital, Edina, Minnesota
  - Mercy and Unity Cancer Center at Unity Hospital, Fridley, Minnesota
  - Hutchinson Area Health Care, Hutchinson, Minnesota
  - Meeker County Memorial Hospital, Lichfield, Minnesota
  - Immanuel St. Joseph's, Mankato, Minnesota
  - HealthEast Cancer Care at St. John's Hospital, Maplewood, Minnesota
  - Minnesota Oncology Hematology, PA - Maplewood, Maplewood, Minnesota
  - Virginia Piper Cancer Institute at Abbott - Northwestern Hospital, Minneapolis, Minnesota
  - Hennepin County Medical Center - Minneapolis, Minneapolis, Minnesota
  - CCOP - Metro-Minnesota, Saint Louis Park, Minnesota
  - HealthEast Cancer Care at St. Joseph's Hospital, Saint Paul, Minnesota
  - United Hospital, Saint Paul, Minnesota
  - St. Francis Cancer Center at St. Francis Medical Center, Shakopee, Minnesota
  - HealthEast Cancer Care at Woodwinds Health Campus, Woodbury, Minnesota
  - Minnesota Oncology Hematology, PA - Woodbury, Woodbury, Minnesota
  - Bismarck Cancer Center, Bismarck, North Dakota
  - Medcenter One Hospital Cancer Care Center, Bismarck, North Dakota
  - Mid Dakota Clinic, PC, Bismarck, North Dakota
  - Adena Regional Medical Center, Chillicothe, Ohio
  - Riverside Methodist Hospital Cancer Care, Columbus, Ohio
  - CCOP - Columbus, Columbus, Ohio
  - Grant Riverside Cancer Services, Columbus, Ohio
  - Mount Carmel Health - West Hospital, Columbus, Ohio
  - Doctors Hospital at Ohio Health, Columbus, Ohio
  - Grady Memorial Hospital, Delaware, Ohio
  - Fairfield Medical Center, Lancaster, Ohio
  - Strecker Cancer Center at Marietta Memorial Hospital, Marietta, Ohio
  - Licking Memorial Cancer Care Program at Licking Memorial Hospital, Newark, Ohio
  - Mercy Medical Center, Springfield, Ohio
  - Community Hospital of Springfield and Clark County, Springfield, Ohio
  - Mount Carmel St. Ann's Cancer Center, Westerville, Ohio
  - Genesis - Good Samaritan Hospital, Zanesville, Ohio
  - Avera Cancer Institute, Sioux Falls, South Dakota
  - Medical X-Ray Center, PC, Sioux Falls, South Dakota
  - Sanford Cancer Center at Sanford USD Medical Center, Sioux Falls, South Dakota

REFERENCES:
- [Result] Kottschade LA, Sloan JA, Mazurczak MA, Johnson DB, Murphy BP, Rowland KM, Smith DA, Berg AR, Stella PJ, Loprinzi CL. The use of vitamin E for the prevention of chemotherapy-induced peripheral neuropathy: results of a randomized phase III clinical trial. Support Care Cancer. 2011 Nov;19(11):1769-77. doi: 10.1007/s00520-010-1018-3. Epub 2010 Oct 9. PMID 20936417

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Two-hundred and seven (207) participants were recruited between December 2006 and December 2007 from 23 North Central Cancer Treatment Group (NCCTG) member sites.
Pre-assignment Details: There were a total of 11 cancellations (4 Vitamin E, 7 Placebo), 1 major violation on Placebo and 7 ineligible (3 Vitamin E and 4 Placebo) participants. Of these, 18 participants of cancellations/ineligible were excluded from all analysis.
Groups:
- Vitamin E: Patients receive oral vitamin E twice daily beginning within 4 days of the start of chemotherapy course 1 and continuing until 1 month after completion of chemotherapy.
- Placebo: Patients receive oral placebo twice daily beginning within 4 days of the start of chemotherapy course 1 and continuing until 1 month after completion of chemotherapy.
Period: Overall Study
Arm/Group | Vitamin E | Placebo
Started | 96 | 93
Completed | 67 | 60
Not Completed | 29 | 33
Not completed — Withdrawal by Subject | 11 | 18
Not completed — Adverse Event | 8 | 3
Not completed — Alternate Treatment | 2 | 4
Not completed — Other Medical Problems | 2 | 4
Not completed — Death | 0 | 1
Not completed — Other Reasons | 6 | 3

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Vitamin E | Placebo | Total
Number analyzed (Participants) | 96 | 93 | 189
Age, Customized [Number; unit: participants]
  <=50 years | 40 | 34 | 74
  >50 years | 56 | 59 | 115
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 80 | 75 | 155
  Male | 16 | 18 | 34
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 2 | 0 | 2
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 2 | 5 | 7
  White | 91 | 87 | 178
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 1 | 1 | 2
Region of Enrollment [Number; unit: participants]
  United States | 96 | 93 | 189
Type of cancer [Number; unit: participants]
  Breast | 58 | 57 | 115
  Lung | 1 | 4 | 5
  Other Cancer | 37 | 32 | 69
Planned number of chemotherapy cycles [Number; unit: participants]
  <=4 | 48 | 49 | 97
  >4 | 48 | 44 | 92
Type of chemotherapy [Number; unit: participants]
  Taxane | 57 | 52 | 109
  Cisplatin | 4 | 4 | 8
  Carboplatin | 1 | 1 | 2
  Oxaliplatin | 24 | 26 | 50
  Combination | 10 | 10 | 20

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Patients With Chemotherapy-induced Sensory Peripheral Neuropathy ≥ Grade 2
Description: The chemotherapy-induced sensory peripheral neuropathy utilized the sensory neuropathy item from the Common Terminology Criteria for Adverse Events (CTCAE) v3.0. Grading: Grade 0=none; grade 1=loss of deep tendon reflexes or paresthesia, including tingling, but not interfering with function; grade 2=objective sensory alteration or paresthesia, including tingling, interfering with function, but not with activities of daily living; grade 3=sensory alteration or paresthesia interfering with activities of daily living; grade 4=permanent sensory losses that are disabling; and grade 5=death.
Time Frame: 6 months post completion of chemotherapy treatment
Population: Participants who received at least one dose of assigned therapy.
Measure: Number; unit: percentage of participants
Arm/Group | Vitamin E | Placebo
Number analyzed (Participants) | 96 | 93
percentage of participants | 34 | 29
Statistical Analysis 1: Comparison: Vitamin E vs Placebo; Test type: Superiority or Other; p = 0.43, Chi-squared

2. Secondary Outcome: Percentage of Patients Requiring Dose Reductions of Chemotherapy Due to Sensory Peripheral Neuropathy
Time Frame: 6 months post completion of chemotherapy treatment
Measure: Number; unit: percentage of patients
Arm/Group | Vitamin E | Placebo
Number analyzed (Participants) | 96 | 93
percentage of patients | 3 | 5
Statistical Analysis 1: Comparison: Vitamin E vs Placebo; Test type: Superiority or Other; p = 0.49, Fisher Exact

3. Secondary Outcome: Percentage of Patients Stopping Chemotherapy Before Treatment is Complete Due to Sensory Peripheral Neuropathy
Time Frame: 6 months post completion of chemotherapy treatment
Measure: Number; unit: percentage of participants
Arm/Group | Vitamin E | Placebo
Number analyzed (Participants) | 96 | 93
percentage of participants | 4 | 3
Statistical Analysis 1: Comparison: Vitamin E vs Placebo; Test type: Superiority or Other; p = 1.00, Fisher Exact

4. Secondary Outcome: Time to Onset of Sensory Peripheral Neuropathy ≥ Grade 2
Description: Time to onset of sensory peripheral neuropathy was calculated using incidences of the adverse event while the patient was receiving chemotherapy.
Time Frame: 6 months post completion of chemotherapy treatment
Measure: Median (95% Confidence Interval); unit: days
Arm/Group | Vitamin E | Placebo
Number analyzed (Participants) | 96 | 93
days | 58 [43 to 97] | 69 [49 to 105]

5. Secondary Outcome: Duration of Sensory Peripheral Neuropathy ≥ Grade 2
Description: Duration of sensory peripheral neuropathy is the time from onset of grade 2+ neuropathy until the neuropathy is resolved to grade 1 or less during chemotherapy treatment.
Time Frame: 6 months post completion of chemotherapy treatment
Measure: Median (95% Confidence Interval); unit: days
Arm/Group | Vitamin E | Placebo
Number analyzed (Participants) | 33 | 27
days | 36 [28 to 44] | NA [NA to NA] — Only 6 participants were resolved before the patient went off study thus median days to resolution and 95% Confidence Interval can not be determined.

ADVERSE EVENTS:
Time Frame: Prior to each cycle of chemotherapy to six months post chemotherapy completion
Arm/Group | Vitamin E | Placebo
Serious Adverse Events (participants affected / at risk) | 0/96 | 0/93
Other Adverse Events (participants affected / at risk) | 26/96 | 25/93
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Vitamin E (N=96) | Placebo (N=93)
Febrile neutropenia (Blood and lymphatic system disorders) | 0 (0) | 2 (2)
Hemoglobin decreased (Blood and lymphatic system disorders) | 1 (1) | 1 (1)
Atrial fibrillation (Cardiac disorders) | 0 (0) | 1 (1)
Tinnitus (Ear and labyrinth disorders) | 1 (1) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 2 (2) | 2 (2)
Constipation (Gastrointestinal disorders) | 0 (0) | 3 (4)
Diarrhea (Gastrointestinal disorders) | 6 (9) | 3 (3)
Esophageal mucositis (Gastrointestinal disorders) | 0 (0) | 1 (1)
Flatulence (Gastrointestinal disorders) | 1 (1) | 0 (0)
Nausea (Gastrointestinal disorders) | 5 (6) | 1 (1)
Vomiting (Gastrointestinal disorders) | 5 (5) | 0 (0)
Edema limbs (General disorders) | 0 (0) | 2 (2)
Fatigue (General disorders) | 2 (3) | 2 (2)
General symptom (General disorders) | 1 (1) | 0 (0)
Hypersensitivity (Immune system disorders) | 1 (1) | 1 (1)
Abdominal infection (Infections and infestations) | 0 (0) | 1 (1)
Pharyngitis (Infections and infestations) | 1 (1) | 0 (0)
Pneumonia (Infections and infestations) | 0 (0) | 1 (1)
Skin infection (Infections and infestations) | 0 (0) | 1 (1)
Upper respiratory infection (Infections and infestations) | 1 (1) | 0 (0)
Urinary tract infection (Infections and infestations) | 1 (1) | 0 (0)
Vascular access complication (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Coagulopathy (Investigations) | 0 (0) | 1 (2)
Leukocyte count decreased (Investigations) | 3 (6) | 2 (2)
Lymphocyte count decreased (Investigations) | 1 (2) | 0 (0)
Neutrophil count decreased (Investigations) | 2 (3) | 4 (6)
Platelet count decreased (Investigations) | 2 (2) | 2 (2)
Anorexia (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Dehydration (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Hyperkalemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Hypoalbuminemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Hypocalcemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Hypokalemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Joint pain (Musculoskeletal and connective tissue disorders) | 2 (6) | 1 (1)
Myalgia (Musculoskeletal and connective tissue disorders) | 2 (5) | 2 (2)
Dizziness (Nervous system disorders) | 1 (1) | 0 (0)
Headache (Nervous system disorders) | 1 (1) | 0 (0)
Intracranial hemorrhage (Nervous system disorders) | 0 (0) | 1 (1)
Ischemia cerebrovascular (Nervous system disorders) | 1 (1) | 0 (0)
Peripheral sensory neuropathy (Nervous system disorders) | 3 (3) | 4 (7)
Syncope (Nervous system disorders) | 1 (1) | 0 (0)
Anxiety (Psychiatric disorders) | 0 (0) | 1 (1)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 3 (3)
Hemorrhage nasal (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Alopecia (Skin and subcutaneous tissue disorders) | 2 (3) | 0 (0)
Hand-and-foot syndrome (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Pruritus (Skin and subcutaneous tissue disorders) | 1 (3) | 0 (0)
Rash desquamating (Skin and subcutaneous tissue disorders) | 1 (1) | 1 (1)
Hemorrhage (Vascular disorders) | 0 (0) | 1 (1)
Hot flashes (Vascular disorders) | 0 (0) | 1 (1)
Hypertension (Vascular disorders) | 0 (0) | 1 (1)
Thrombosis (Vascular disorders) | 0 (0) | 5 (5)
Visceral arterial ischemia (Vascular disorders) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes